CLINICAL TRIAL: NCT03755778
Title: A Non-Randomized, Open-Label, Three-Part, Drug-Drug Interaction Study to Evaluate the Effects of Itraconazole, Rifampin, and Quinidine on the Pharmacokinetics and Safety of EDP-938 in Healthy Subjects
Brief Title: Drug-Drug Interaction Study Between EDP-938, Itraconazole, Rifampin, and Quinidine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: Pharmaceutical Research Associates (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EDP 938-003
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2018-10

CONDITIONS: RSV Infection
Keywords: drug-drug interaction
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — EDP-938; Itraconazole; Rifampin; Quinidine

STUDY DESIGN:
Intervention Model Description: 3-Part Single Group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EDP-938 and itraconazole interaction (Part 1) (Experimental)
  Interventions: Drug: EDP-938; Drug: Itraconazole
- EDP-938 and rifampin interaction (Part 2) (Experimental)
  Interventions: Drug: EDP-938; Drug: Rifampin
- EDP-938 and quinidine interaction (Part 3) (Experimental)
  Interventions: Drug: EDP-938; Drug: Quinidine

INTERVENTIONS:
Drug: EDP-938 — Subjects will receive EDP-938 once daily on Day 1 and 14 (Part 1)
  Arms: EDP-938 and itraconazole interaction (Part 1)
Drug: EDP-938 — Subjects will receive EDP-938 once daily on Day 1 and 14 (Part 2)
  Arms: EDP-938 and rifampin interaction (Part 2)
Drug: EDP-938 — Subjects will receive EDP-938 once daily on Day 1 and 8 (Part 3)
  Arms: EDP-938 and quinidine interaction (Part 3)
Drug: Itraconazole — Subjects will receive itraconazole once daily from Day 5 to Day 18
  Arms: EDP-938 and itraconazole interaction (Part 1)
Drug: Rifampin — Subjects will receive rifampin once daily from Day 5 to Day 16
  Arms: EDP-938 and rifampin interaction (Part 2)
Drug: Quinidine — Subjects will receive quinidine once daily from Day 5 to Day 12
  Arms: EDP-938 and quinidine interaction (Part 3)

SUMMARY:
A Non-Randomized, Open-Label, Three-Part, Drug-Drug Interaction Study to Evaluate the Effects of Itraconazole, Rifampin, and Quinidine on the Pharmacokinetics and Safety of EDP-938 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 55 years, inclusive.
* Screening body mass index (BMI) of 18 to 30 kg/m2 with a minimum body weight of 50 kg
* Female subjects of childbearing potential must agree to use two effective methods of contraception from the date of Screening until 90 days after the last dose of EDP 938.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease.
* For Part 3 subjects, the following cardiovascular abnormalities:

  * QRS duration >110 ms
  * Incomplete right bundle branch block or any complete bundle branch block
  * Heart rate <40 or >90 beats per minute (per vital sign capture while rested)
  * History of unexplained syncope, structural heart disease, or clinically significant arrhythmias
  * Personal or family history of long QT syndrome (genetically proven or suggested by sudden death of a close relative due to cardiac causes at a young age) or Brugada syndrome
  * PR interval >220 ms or any 2nd or 3rd degree AV block
  * Ventricular pre-excitation
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at Screening or Day -1.
* Current tobacco smokers or use of tobacco within 3 months prior to Screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of regular alcohol consumption.
* Participation in a clinical trial within 30 days prior to the first dose of study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-27 (Actual)

PRIMARY OUTCOMES:
Cmax of EDP-938 with and without coadministration with itraconazole | Up to 19 days
AUC of EDP-938 with and without coadministration with itraconazole | Up to 19 days
Cmax of EDP-938 with and without coadministration with rifampin | Up to 17 days
AUC of EDP-938 with and without coadministration with rifampin | Up to 17 days
Cmax of EDP-938 with and without coadministration with quinidine | Up to 13 days
AUC of EDP-938 with and without coadministration with quinidine | Up to 13 days

SECONDARY OUTCOMES:
Safety measured by adverse events | Up to 25 days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- Pharmaceutical Research Associates, Inc.,, Lenexa, Kansas, United States